CLINICAL TRIAL: NCT05638555
Title: Lactated Ringers vs Normal Saline in Patients With Acute Pancreatitis: A Bias-Adjusted Meta-analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qatar University (Other)
Responsible Party: Principal Investigator, Yaman Khamis, Group Leader, Qatar University
Other Study IDs: 1983542-1
Record Dates: First submitted 2022-11-13; First posted 2022-12-06 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lactated Ringer's (LR) solution
- Normal Saline (NS)

SUMMARY:
This study aims to compare NS and LR in terms of outcomes in patients with acute pancreatitis while addressing the current methodological issues with available meta-analyses on the topic. Such comparison combined with bias adjustment will assist with identifying the optimal fluid rehydration therapy in acute pancreatitis, since most of the available data is conflicted around the topic. A database search will be conducted to identify studies comparing normal saline and ringer's lactate. Existing meta-analyses will be assessed. The results will be discussed in the light of their strengths and limitations and then any deficiencies will be addressed through a new synthesis as a final step of this umbrella review. The primary outcome will be SIRS at 24 hours. OR and 95% confidence intervals will be generated using the quality effects model. Heterogeneity will be evaluated using the I2 statistic. Publication bias will be assessed using the Doi Plot.

ELIGIBILITY:
Inclusion Criteria:

* RCTs and observational studies that compared NS vs LR in AP patients.
* Studies reviewed must report data as effect estimates or provide raw data sufficient to calculate effect estimates.

Exclusion Criteria:

* Studies involving animal studies, pediatric patient populations, and cell lines will be excluded.

All studies will be reviewed in full form by each author to determine eligibility. In case of disagreement, determination of inclusion will be reached via consensus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult Patients diagnosed with Acute Pancreatitis (AP)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Systemic inflammatory response syndrome (SIRS) | at 24 hours
  SIRS is defined as two out of the following four criteria:
  a) Temperature<36˚C (96.8˚F) or >38˚C (100.4˚F) b) Heart rate>90/min c) Respiratory rate>20/min d) WBC(<4000/mm3) (>12,000/mm3) or 10% bands.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Doi, Principal Investigator — Qatar University
Locations (1):
- Suhail Doi, Doha, Qatar